CLINICAL TRIAL: NCT02762032
Title: The Ability of an Oral Supplement to Improve Skin Microperfusion, Hydration, Elasticity, and Barrier Function
Brief Title: Natreon Healthy Skin Study - PrimaVie Supplement
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Collaborators: Natreon, Inc. (Industry)
Responsible Party: Principal Investigator, Gayle Gordillo, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DCS-71-14
Record Dates: First submitted 2016-03-21; First posted 2016-05-04 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: Skin Biopsy; PrimaVie; Herbal Supplement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): 15 subjects will be randomized to receive PrimaVie Herbal Supplement 125 mg to take twice daily for 14 weeks.
  Interventions: Dietary Supplement: PrimaVie Herbal Supplement 125
- Arm 2 (Active Comparator): 15 subjects will be randomized to receive PrimaVie Herbal Supplement 250 mg to take twice daily for 14 weeks.
  Interventions: Dietary Supplement: PrimaVie Herbal Supplement 250
- Arm 3 (Placebo Comparator): 15 subjects will be randomized to receive placebo (control supplement) to take twice daily for 14 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: PrimaVie Herbal Supplement 125 — 125 mg to take BID for 14 weeks in Arm 1
  Other Names: PrimaVie
  Arms: Arm 1
Dietary Supplement: PrimaVie Herbal Supplement 250 — 250 mg to take BID for 14 weeks in Arm 2
  Other Names: PrimaVie
  Arms: Arm 2
Drug: Placebo — Placebo supplement to take BID for 14 weeks in Arm 3
  Other Names: control supplement
  Arms: Arm 3

SUMMARY:
This study will demonstrate the ability of the oral supplement, PrimaVie® to improve skin microperfusion, hydration, elasticity and barrier function. 45 females will be enrolled in 1 of 3 arms where they will receive either 125 mg PrimaVie, 250 mg PrimaVie or placebo (control) to take twice daily for 14 weeks.

DETAILED DESCRIPTION:
Subjects will be assessed based on they type of Fitzpatrick skin type they have, will be return for a total of 6 study visits over 14 weeks where the following research activities will take place through the course of the study: medical/dietary history, medications will be recorded, supplement randomization based on one of the three arms will occur at study visit 1, and distribution of the study product will occur at all study visits, supplement tolerabiltity assessment, investigator and subject appearance assessment, photography of the face (left, right and front) will be taken, non-invasive assessments including Trans-epidermal Water Loss, hydration, elasticity, laser speckle perfusion, a skin biopsy of left inner upper arm (only at study visits 2 and 6), adverse event review, and supplement count/compliance review.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to discontinue any dietary or nutritional supplements, other than a general multivitamin, starting two weeks before onset of study and also during the study.
* Subjects must be willing to maintain their present diet with no major changes throughout the study.
* Subjects must be willing to take the dietary supplements as required by the study protocol twice daily.
* Female subjects must be between the ages of 30 to 65 years of age
* Subjects must provide written informed consent and are willing to comply with all study procedures.

Exclusion Criteria:

* Any dermatological disorder that may interfere with the accurate evaluation of the subject's skin.
* Subjects who are pregnant, breast feeding, or planning a pregnancy.
* Clinically significant unstable medical disorders.
* History of, diabetes, heart or kidney disease
* History of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
* Any skin disease in the area of the upper inner arm where the biopsies will be obtained.
* Currently taking the following medications:

  * Steroids
  * Beta-blockers
  * Immunosuppressant's
  * Hydochlorothiazide,
  * Statins
  * Aspirin
  * ACE Inhibitors
  * Muscle relaxants
  * Stimulants
* Prisoners
* Males

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in non-invasive skin assessment of skin microperfusion | 14 weeks after oral supplementation
  To see the improvement in noninvasive skin assessment of objective measurements such as skin microperfusion (laser speckle contrast imaging) (scale Pu)
Improvement in non-invasive skin assessment of hydration | 14 weeks after oral supplementation
  To see the improvement in noninvasive skin assessment of objective measurements such as skin hydration using the DermaLab Combo Series (unit of micro-Siemens uS)
Improvement in non-invasive skin assessment of elasticity | 14 weeks after oral supplementation
  To see the improvement in noninvasive skin assessment of objective measurements such as skin elasticity using the DermaLab Combo Series (mega Pascal mPa and ms units)
Improvement in non-invasive skin assessment of barrier function | 14 weeks after oral supplementation
  To see the improvement in noninvasive skin assessment of objective measurements such as barrier function using Trans-Epidermal Water Loss using the DermaLab Combo Series (g/m2/h)

SECONDARY OUTCOMES:
Gene Chip Analysis | 14 weeks
  identify the up or down regulation of key youthful skin markers (gene expression) produced by the supplement over the placebo as identified by gene chip analysis after 14 weeks of oral supplementation.

OTHER OUTCOMES:
Subjective visual assessment by photographs | 14 weeks
  Identify subjectively by visual assessment, the effect of the PrimaVie supplement on skin appearance by the investigator/study physician at the end of 14 weeks of treatment from photographs taken at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M Gordillo, M.D., Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - OSU Hospital East, Columbus, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Martha Morehouse Medical Plaza 2050 Kenny Road, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das A, S El Masry M, Gnyawali SC, Ghatak S, Singh K, Stewart R, Lewis M, Saha A, Gordillo G, Khanna S. Skin Transcriptome of Middle-Aged Women Supplemented With Natural Herbo-mineral Shilajit Shows Induction of Microvascular and Extracellular Matrix Mechanisms. J Am Coll Nutr. 2019 Aug;38(6):526-536. doi: 10.1080/07315724.2018.1564088. Epub 2019 Jun 4. PMID 31161927